CLINICAL TRIAL: NCT04635189
Title: A Phase II Study of Steroid Sparing Treatment With Daratumumab and Lenalidomide in Newly Diagnosed Transplant Ineligible Patients With Multiple Myeloma
Brief Title: Steroid Sparing Treatment With in Newly Diagnosed Transplant Ineligible Patients With Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Frank Passero, Professor of Hematology/Oncology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMMY20033
Record Dates: First submitted 2020-11-12; First posted 2020-11-19 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental Arm: Cycle 1-4 All subjects (Active Comparator): Subjects will be treated with the following:
  * Daratumumab 16 milligrams/kilograms intravenously weekly for 8 treatments, followed by every 2 weeks for 8 treatments, followed by every 4 weeks
  * Lenalidomide 25 milligrams by mouth daily days 1-21 out of a 28 day cycle
  * Dexamethasone 20 milligrams by mouth or intravenously at least 60 minutes prior to first infusion of daratumumab
  Interventions: Drug: Daratumumab; Drug: Lenalidomide; Drug: Dexamethasone
- Experimental Arm: Cycle 5+ Partial Response or Better (Experimental): Subjects will be treated the following:
  * Daratumumab 16 milligrams/kilograms intravenously weekly for 8 treatments, followed by every 2 weeks for 8 treatments, followed by every 4 weeks
  * Lenalidomide 25 milligrams/kilograms daily days 1-21 out of a 28 day cycle
  Interventions: Drug: Daratumumab; Drug: Lenalidomide
- Experimental Arm: Cycle 5+ Less than Partial Response (Active Comparator): Subjects will be treated the following:
  * Daratumumab 16 milligrams/kilograms intravenously weekly for 8 treatments, followed by every 2 weeks for 8 treatments, followed by every 4 weeks
  * Lenalidomide 25 milligrams by mouth daily days 1-21 out of a 28 day cycle
  * Dexamethasone 20 milligrams by mouth or intravenously at least 60 minutes prior to first infusion of daratumumab
  Interventions: Drug: Daratumumab; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Daratumumab 16 milligrams/kilograms intravenously weekly for 8 treatments, followed by every 2 weeks for 8 treatments, followed by every 4 weeks
  Other Names: Darzalex
Drug: Lenalidomide — Lenalidomide 25 milligrams by mouth daily days 1-21 out of a 28 day cycle
  Other Names: Revlimid
Drug: Dexamethasone — Dexamethasone 20 milligrams by mouth or intravenously at least 60 minutes prior to first infusion of daratumumab
  Other Names: Ozurdex
  Arms: Experimental Arm: Cycle 1-4 All subjects; Experimental Arm: Cycle 5+ Less than Partial Response

SUMMARY:
The purpose of this study is to determine the effects of daratumumab and lenalidomide without steroids for treating patients with multiple myeloma.

DETAILED DESCRIPTION:
This is an open label, phase 2 study consisting of daratumumab, lenalidomide and dexamethasone, given upfront in newly diagnosed, transplant ineligible patients with myeloma. Patients participating in the study will be recruited from the Wilmot Cancer Institute, University of Rochester in Rochester, New York and all University of Rochester community affiliates.

Patients will be treated with 1800 milligrams of Daratumumab subcutaneously or 16 milligrams/kilograms daratumumab intravenously (IV) weekly for 8 treatments, followed by every 2 weeks for 8 treatments, followed by every 4 weeks. Patients will be treated with 25 milligrams of Lenalidomide days 1-21 out of a 28 day cycle (dose adjustments for creatinine clearance) and 20 milligrams of Dexamethasone at least 60 minutes prior to first infusion of daratumumab. Each cycle consists of 28 days (4 weeks).

Response assessments by International Myeloma Working Group criteria for myeloma will be performed every 4 weeks while on therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma with diagnosis
* Must not have received previous therapy for multiple myeloma
* Newly diagnosed and not considered candidate for high-dose chemotherapy
* Adequate organ system function
* A performance status ≤ 3
* Ability to swallow and retain oral medication
* Female subjects of child bearing potential must be surgically sterile, be post-menopausal

Exclusion Criteria:

* A diagnosis of primary amyloidosis; monoclonal gammopathy of undetermined significance, smoldering multiple myeloma; non-secretory myeloma
* A diagnosis of Waldenström's disease
* Receiving cancer therapy
* Radiation therapy within 14 days of enrollment
* Major surgery within 2 weeks before enrollment
* Human immunodeficiency virus -infected patients must be on effective anti-retroviral therapy with undetectable viral load within the past 6 months
* Seropositive for hepatitis B, or seropositive for hepatitis C
* Ongoing systemic bacterial, fungal or viral infection
* Severe and/or uncontrolled medical conditions
* Malignancy within 2 years of study enrollment
* Women who are pregnant or lactating
* Contraindications to required prophylaxis for deep vein thrombosis and pulmonary embolism.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Daratumumab Related Infusion Reactions | 28 days
  To determine the rate of daratumumab related infusion reactions in patients treated for myeloma without steroids compared to historical controls.

SECONDARY OUTCOMES:
Determination of Response Rates | 28 days
  To determine the proportion of patients who do not achieve at least a partial response after 4 cycles and require steroids to be added back to their regimen

CONTACTS AND LOCATIONS:
Overall Officials: Frank Passero, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial will be shared after deidentification, including dictionaries.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data for any type of analyses.